CLINICAL TRIAL: NCT02968511
Title: EGESTA - Emergent GI Therapy for Severe, Complicated CDI Using Fecal Microbiota
Brief Title: EGESTA - Emergent GI Therapy for Severe, Complicated CDI Using Fecal Microbiota Transplant
Acronym: EGESTA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible patients
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: OpenBiome (Industry)
Responsible Party: Principal Investigator, David B. Stewart, MD, FACS, FASCRS, Associate Professor of Surger, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005388
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: C.Difficile Colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fecal microbiota transplant (Experimental): 250 mL of fecal transplant material by enema as treatment
  Interventions: Biological: fecal microbiota transplant

INTERVENTIONS:
Biological: fecal microbiota transplant — Fecal microbiota transplant for the treatment of severe, complicated C. difficile infection
  Other Names: FMT Microbiota Preparation

SUMMARY:
The objectives/specific aims of this study are three-fold. First, the study seeks to evaluate the safety of fecal microbiota transplant (FMT) in patients with severe, complicated C. difficile infection (scCDI). Second, the study seeks to evaluate whether fecal microbiota transplant (FMT) can improve scCDI, with "improve" defined as either decreasing the severity of CDI, or by resolving the infection altogether. Third, the study seeks to further study the mechanism by which FMT improves the course of scCDI by performing 16S rRNA and ITS sequencing on pre-FMT and serial post-FMT stool samples in order to measure changes to bacterial and fungal microbiota as a consequence of CDI and FMT therapy. FMT material (hereafter referred to as FMTm) would be obtained from OpenBiome. FMTm is prepared from prescreened healthy donors.

The hypothesis of the study is that FMT is a preferred salvage therapy for scCDI as compared to (1) ongoing, failing medical therapy with conventional antibiotics and (2) surgery.

DETAILED DESCRIPTION:
The objectives/specific aims of this study are three-fold. First, the study seeks to evaluate the safety of fecal microbiota transplant (FMT) in patients with severe, complicated C. difficile infection (scCDI). Second, the study seeks to evaluate whether fecal microbiota transplant (FMT) can improve scCDI, with "improve" defined as either decreasing the severity of CDI, or by resolving the infection altogether. Third, the study seeks to further study the mechanism by which FMT improves the course of scCDI by performing 16S rRNA and ITS sequencing on pre-FMT and serial post-FMT stool samples in order to measure changes to bacterial and fungal microbiota as a consequence of CDI and FMT therapy. FMT material (hereafter referred to as FMTm) would be obtained from OpenBiome. FMTm is prepared from prescreened healthy donors.

The hypothesis of the study is that FMT is a preferred salvage therapy for scCDI as compared to (1) ongoing, failing medical therapy with conventional antibiotics and (2) surgery.

The standard of care treatment for scCDI is conventional antibiotics with either parenteral/oral metronidazole, and/or vancomycin provided in the form of oral and/or retention enemas. The reliability of these conventional antibiotics in the setting of scCDI is very unpredictable, and patients with CDI of this severity have a mortality rate that in some series is greater than 50%. It is against the mediocre historical record of these antibiotics that FMT would be tested in this highly moribund patient population.

FMT would not be provided to patients with scCDI off protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 years of age and 75 years of age.
* Have CDI defined as clinical symptoms of CDI (diarrhea with or without abdominal pain/abdominal distention) with a confirmatory nucleic acid amplification test (NAAT) positive for CDI.
* Have severe/complicated disease as defined by ACG guidelines(appendix 1), with any of the following attributable to CDI:

  * Admission to intensive care unit for CDI
  * Hypotension (systolic blood pressure < 90 mmHg) with or without required use of vasopressors
  * Fever ≥ 38.5 ° C
  * Ileus (as defined by the absence of intestinal function for at least 24 hours and/or radiographic evidence of pathologically dilated small intestine without evidence of a mechanical obstruction) or significant abdominal distention
  * Mental status changes
  * WBC ≥ 35,000 cells / mm 3 or < 2,000 cells / mm 3
  * Serum lactate levels >2.2 mmol / l
  * End organ failure (mechanical ventilation,renal failure as defined by a rise in creatinine of >1.5 mg/dL either above the upper limit of normal for creatinine, or > 1.5 mg/dL from premorbid levels if that information is known, acute hepatic dysfunction as defined by an increase in AST or ALT to twice the upper limit of normal, etc.)

Exclusion Criteria:

* Pregnant or lactating women
* Prisoners
* Patients under the age of 18 or over the age of 76 years of age
* Patients who are immunocompromised including but not limited to:

  * Have HIV infection historically reported, regardless of CD4 count
  * AIDS as defined by either an AIDS-defining diagnosis (appendix 2) or a CD4 count <200/mm3,
  * Inherited or primary immune disorders,
  * Received chemotherapy within the previous 90 days, or
  * Current or recent treatment with any immunosuppressant medications in the past 90 days
* Individuals who have received FMT at any time before potential study enrollment
* Patients who do not have a stool test confirming C. difficile infection
* Patients who have a severe anaphylactic response to food
* Patients with allergies to sodium chloride or glycerol, both ingredients Generally Recognized As Safe (GRAS)
* Patients who have colorectal cancer
* Diagnosis of Irritable Bowel Disease or Irritable Bowel Syndrome
* Any other condition for which the Principal Investigator thinks the treatment may pose a health risk
* Anticipated or predicted death within the time period of follow-up for reasons unrelated to CDI
* An APACHE II score >29 at the time of evaluation for inclusion in the study protocol (Appendix 4.0)
* Mandatory ongoing antibiotic use for non-CDI infection
* Patients unable to provide informed consent or who do not have a legally authorized representative for consent
* Patients unable to comply with requirements of this study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Safety - adverse events | Thirty days after treatment
  Absence of unexpected related adverse events

SECONDARY OUTCOMES:
Efficacy (Cure of infection, or decrease in severity of infection based on white blood cell count) | Thirty days after treatment
  Cure of infection, or decrease in severity of infection based on white blood cell count

CONTACTS AND LOCATIONS:
Locations (1):
- David Stewart, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No